CLINICAL TRIAL: NCT02475265
Title: Transdermal Estrogen in Older Premenopausal Women With Anorexia Nervosa
Acronym: 1180
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Pouneh K. Fazeli, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P000463; R03DK106410 (NIH)
Record Dates: First submitted 2015-06-10; First posted 2015-06-18 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Anorexia Nervosa; Osteoporosis
Keywords: Anorexia Nervosa; Osteoporosis; Eating Disorder; Disordered Eating; Estrogen; Bone
MeSH Terms: conditions — Anorexia Nervosa; Osteoporosis; Feeding and Eating Disorders | interventions — Estradiol; Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- estradiol 0.045mg/levonorgestrel 0.015mg (Experimental): 6 months of estradiol 0.045mg/levonorgestrel 0.015mg (once weekly patch).
  Interventions: Drug: estradiol 0.045 mg/levonorgestrel 0.015mg

INTERVENTIONS:
Drug: estradiol 0.045 mg/levonorgestrel 0.015mg
  Other Names: Climara Pro transdermal patch

SUMMARY:
Decreased bone strength is a common and serious medical problem present in many women with anorexia nervosa. Women with decreased bone strength are more likely to suffer broken bones than women with normal bone strength.

This study will investigate whether the use of transdermal estrogen can improve bone mineral density (BMD) and bone microarchitecture in women with anorexia nervosa anorexia nervosa when used for 6 months.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a prevalent psychiatric disorder affecting up to 1% of college-aged women in the US and an increasing number of women over 30 years of age. Among the many medical co-morbidities associated with AN, the most common is significant bone loss, which can persist despite weight recovery. Nearly 50% of women with AN have osteopenia with an additional 30% meeting WHO criteria for osteoporosis. Importantly, this severe bone loss is associated with an increased fracture risk. Nearly 30% of women with AN report a history of a fracture and a prospective study demonstrated a 7-fold increased risk of fracture in women with AN compared to age-matched controls. Because AN is a chronic disease that can persist despite psychiatric and nutritional counseling, the bone loss and increased fracture risk can persist and lead to lifelong morbidity. Therefore, finding a treatment for bone loss associated with AN is of critical importance.

This 6 month open-label study will investigate in women (ages 25 to 50 years old) with AN whether treatment with transdermal estrogen replacement will increase bone mineral density (BMD), improve parameters of bone microarchitecture as assessed by high-resolution peripheral quantitative computed tomography (HR-pQCT), and improve bone strength as estimated by microfinite element analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female; ages 25-50 years
* Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) psychiatric criteria for AN, including <85% of ideal body weight as defined by the 1983 Metropolitan Life Insurance Height and Weight Tables, and amenorrhea
* T-score of < -1.5 at spine or hip
* Treatment team or treatment professional in place for clinical treatment/monitoring during the study

Exclusion Criteria:

* Diseases known to affect bone metabolism, including untreated thyroid dysfunction, vitamin D deficiency, Cushing's syndrome, diabetes mellitus or renal insufficiency
* Personal history of venous or arterial clot
* History of stroke or myocardial infarction
* History of migraine headaches
* History of hypercoagulable disorder
* Personal history or history of a first-degree relative with breast cancer
* History of hereditary angioedema
* Any medication known to affect bone metabolism, including systemic glucocorticoids within three months of the baseline visit, depot medroxyprogesterone within 6 months of the baseline visit, oral bisphosphonates within one year of the baseline visit or intravenous (IV) bisphosphonates within three years of the baseline visit
* Bone fracture within the prior 12 months
* Serum potassium < 3.0 meq/L or serum alanine aminotransferase (ALT) > 3 times the upper limit of normal
* Fasting serum triglyceride level > 150 mg/dL
* Pregnant or breastfeeding
* Active substance abuse

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pouneh K Fazeli, MD, Principal Investigator — MGH/Harvard Medical School
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Estradiol 0.045mg/Levonorgestrel 0.015mg: 6 months of estradiol 0.045mg/levonorgestrel 0.015mg (once weekly patch).
  estradiol 0.045 mg/levonorgestrel 0.015mg
Period: Overall Study
Arm/Group | Estradiol 0.045mg/Levonorgestrel 0.015mg
Started | 11
Completed | 8
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Estradiol 0.045mg/Levonorgestrel 0.015mg
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Lumbar spine bone mineral density [Mean (Standard Deviation); unit: g/cm^2] | 0.776 (0.104)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Bone Mineral Density (BMD) of Lumbar Spine by Dual Energy X-ray Absorptiometry (DXA)
Description: Percent change in lumbar spine bone mineral density after six-months. Lumbar spine bone mineral density measured by dual energy x-ray absorptiometry.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Estradiol 0.045mg/Levonorgestrel 0.015mg
Number analyzed (Participants) | 8
percent change | 2.0 (0.8)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Estradiol 0.045mg/Levonorgestrel 0.015mg
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 7/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Estradiol 0.045mg/Levonorgestrel 0.015mg (N=11)
Nausea (Gastrointestinal disorders) | 3
Breast tenderness (Reproductive system and breast disorders) | 1
Patch site irritation (Skin and subcutaneous tissue disorders) | 3
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT02475265/Prot_SAP_000.pdf